CLINICAL TRIAL: NCT05464849
Title: Evaluation of Systemic Microvascular Reactivity in Patients With Resistant Hypertension
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CAAE 53946021.8.0000.5272
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Arterial Hypertension; Resistant Hypertension; Microvascular Rarefaction; Endothelial Dysfunction
MeSH Terms: conditions — Hypertension; Microvascular Rarefaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Resistant hypertension: Patients presenting with resistant hypertension
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function
- non-resistant hypertension: Patients presenting with non-resistant hypertension
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function
- normotensive subjects: control group including normotensive volunteers
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function

INTERVENTIONS:
Diagnostic Test: Evaluation of systemic skin microvascular endothelial function — Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.

SUMMARY:
Systemic arterial hypertension is a serious health problem worldwide. In some cases, it can phenotypically present as resistant arterial hypertension, which consists of blood pressure levels outside the treatment goals in patients using three or more classes of antihypertensive drugs, one of which is preferably a thiazide diuretic. Resistant hypertension contributes to a 47% higher risk of developing cardiovascular events when compared to patients with non-resistant hypertension. It is known that the microcirculation plays a relevant role in the pathophysiology of arterial hypertension. Furthermore, it is known that the cutaneous microvascular network is an adequate model and that it reflects the systemic microcirculation. In this sense, the present research proposes the study of cutaneous capillary density - through high resolution intravital microscopy - and of the endothelium-dependent and independent microvascular vasodilator response - by the speckle laser flowmetry method coupled to a pharmacological system of micro- iontophoresis - in patients diagnosed with resistant hypertension, with the aim of identifying changes in comparison with patients with non-resistant hypertension and normotensive individuals. Additionally, the evaluation of the association between systemic microvascular function and the presence of target organ lesions in this population may indicate that this is a new non-invasive way of stratifying cardiovascular risk in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension

Exclusion Criteria:

* Pregnancy or lactation for all groups.
* For the control group: endocrine and metabolic diseases, including diabetes mellitus, cardiovascular diseases, including hypertension, autoimmune diseases and cancer.
* For the resistant arterial hypertension and non-resistant arterial hypertension groups: endocrine diseases, except diabetes mellitus, autoimmune diseases and cancer .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Resistant hypertension: Blood pressure levels outside the treatment goals in patients using three or more classes of antihypertensive drugs, one of which is preferably a thiazide diuretic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Systemic microvascular reactivity | two years - during one visit to the microcirculation laboratory
  evaluation of endothelium-dependent and -independent microvascular function

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Tibiriçá, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crahim V, Verri V, De Lorenzo A, Tibirica E. Reduced systemic microvascular function in patients with resistant hypertension and microalbuminuria: an observational study. J Hum Hypertens. 2024 Dec;38(12):806-813. doi: 10.1038/s41371-024-00958-7. Epub 2024 Sep 17. PMID 39289473